CLINICAL TRIAL: NCT03934645
Title: Comparison of Efficacy of "Pre-deliric Version 1-2, E-predeliric Score and ICDSC" Tests Used in the Diagnosis of Delirium in Intensive Care Patients
Brief Title: Comparison of Delirium Evaluation Tools Effectiveness in Intensive Care Patients
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Onur Kucuk, Department of anesthesiology and reanimation Resident Doctor, Trakya University
Other Study IDs: TÜTF-BAEK 2017/263
Record Dates: First submitted 2019-04-19; First posted 2019-05-02 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Delirium
Keywords: delirium; Intensive Care Delirium Screening Checklist (ICDSC); intensive care unit (ICU); Delirium prediction model for ICU patients version 1; Delirium prediction model for ICU patients version 2; Early prediction model for delirium in ICU patients; sensitivity; specificity
MeSH Terms: conditions — Delirium; Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Not In Delirium: Intensive Care Delirium Screening Checklist(ICDSC)=0
  Interventions: Other: Delirium prediction model for ICU patients, version 1; Other: Delirium prediction model for ICU patients, version 2; Other: Early prediction model for delirium in ICU patients
- In Delirium: Intensive Care Delirium Screening Checklist(ICDSC)≥4
  Interventions: Other: Delirium prediction model for ICU patients, version 1; Other: Delirium prediction model for ICU patients, version 2; Other: Early prediction model for delirium in ICU patients

INTERVENTIONS:
Other: Delirium prediction model for ICU patients, version 1 — The pre-deliric model version 1 for intensive care patients consists of ten risk factors that are readily available within 24 hours after intensive care admission and has a high predictive value. The model allows for early prediction of delirium and initiation of preventive measures. Data of the patient in the first 24 hours of admission to the intensive care unit are collected and the delirium prediction score is found.
  Other Names: Pre-deliric version-1
Other: Delirium prediction model for ICU patients, version 2 — The pre-deliric model version 2 for intensive care patients consists of ten risk factors that are readily available within 24 hours after intensive care admission. Data of the patient in the first 24 hours of admission to the intensive care unit are collected and the delirium prediction score is found. The model allows for early prediction of delirium and initiation of preventive measures.
  Other Names: Pre-deliric version-2
Other: Early prediction model for delirium in ICU patients — The e-pre-deliric model enables the clinician to identify those patients likely to develop delirium following ICU admission using only nine predictors. In the e-pre-deliric model, delirium prediction score is determined by inputting the data of the patient in admission to the intensive care unit.
  Other Names: E-pre-deliric

SUMMARY:
This study compares the efficacy of scoring models used in delirium prediction in patients applying to intensive care unit. The diagnosis of delirium is based on the Intensive Care Delirium Screening Checklist (ICDSC). The aim of this study is determine the sensitivity and specificity of three prediction models (Delirium prediction model for ICU patients version 1 [Predeliric version-1], Delirium prediction model for ICU patients version 2 [Predeliric version-2] and Early prediction model for delirium in ICU patients [E-Predeliric]).

DETAILED DESCRIPTION:
Most patients in the intensive care unit (ICU) are entered delirium during hospitalization. Delirium; has been reported that it is associated with significant side effects such as prolonged stay in hospital and intensive care unit, increased morbidity and mortality and high costs. For evaluating delirium in intensive care units; There are several assessment tools such as the Intensive Care Delirium Screening Checklist(ICDSC) etc. The ICDSC checklist is an eight-item screening tool that is based on DSM criteria and applied with data that can be collected through medical records. Its validity has been confirmed by several studies. Assessment tools such as ICDSC; can diagnose after patient is entered the delirium and therefore cannot provide early treatment and preventive measures. Prevention of delirium is more important than the correct treatment of delirium. For preventing delirium; early diagnosis and treatment are necessary. Pre-deliric (DELIRIUM PREDICTION MODEL FOR INTENSIVE CARE PATIENTS) and E-pre-deliric (EARLY PREDICTION MODEL FOR DELIRIUM IN ICU PATIENTS) prediction models; are developed and approved for delirium estimation in intensive care unit patients.

Data of the patient in the first 24 hours of admission to the intensive care unit are collected and the delirium prediction score is found by the pre-deliric model. In the e-pre-deliric model, delirium prediction score is determined by inputting the data of the patient in admission to the intensive care unit.

In this study; the definition of delirium was done by ICDSC scoring. Patients with an ICDSC score of 4 and over were diagnosed with delirium.

The aim of this study; To determine the sensitivity and specificity of E-pre-deliric and Pre-deliric scores by comparing the effectiveness of ICDSC, E-pre-deliric, Pre-deliric version-1 and Pre-deliric version-2 assessment tools in the prediction of delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the intensive care unit for more than 24 hours
* Patients 18 years and older
* Patients without mental disability
* Non-pregnant patients

Exclusion Criteria:

* Patients hospitalized in the intensive care unit for less than 24 hours
* Patients under 18 years
* Patients in coma during hospitalization in the intensive care unit
* Patients with aphasia disease, who cannot communicate
* If the compliance rate of the delirium screening was <%80 during a patient's stay in the ICU
* If signs of delirium are seen within 24 hours of ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In our study, 250 patients hospitalized more than twenty-four hours in the anesthesia intensive care unit of Trakya University Medical Faculty between 01 November 2017 and 01 November 2019 were accepted.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Rate of Predeliric version-1 model | 1 day in admission (1 time)
  Data of the patient (ten risk factors) in the first 24 hours of admission to the intensive care unit are collected and the delirium prediction score is calculated. Each item is scored 0-100.
Rate of Predeliric version-2 model | 1 day in admission (1 time)
  Data of the patient (ten risk factors) in the first 24 hours of admission to the intensive care unit are collected and the delirium prediction score is calculated. Each item is scored 0-100.
Rate of E-predeliric model | 1 day in admission (1 time)
  In the e-pre-deliric model, delirium prediction score is calculated by inputting the data of the patient (nine predictors) in admission to the intensive care unit. Each item is scored 0-100.

SECONDARY OUTCOMES:
ICDSC score | 1 time per day during hospitalization
  The items include the assessment of: (1) consciousness ( deep sedation/coma, agitation, normal wakefulness, or light sedation); (2) inattention; (3) disorientation; (4) hallucination, delusion, or psychosis; (5) psychomotor agitation or retardation; (6) inappropriate speech or mood; (7) sleep-wake cycle disturbances; and (8) fluctuation of symptomatology. The maximum score is eight; scores of ≥4 indicate the presence of delirium and score zero is indicate not in delirium. Each item is scored 0-8.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK MEMİŞ, Proffesor, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Centrum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No